CLINICAL TRIAL: NCT02478645
Title: Dose-ranging Study of Ramosetron for the Prevention of Nausea and Vomiting After Gynecologic Laparoscopic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 4-2014-1065
Record Dates: First submitted 2015-06-18; First posted 2015-06-23 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- ramosetron 0.3 (Experimental)
  Interventions: Drug: ramosetron 0.3
- ramosetron 0.45 (Active Comparator)
  Interventions: Drug: ramosetron 0.45
- ramosetron 0.6 (Active Comparator)
  Interventions: Drug: ramosetron 0.6

INTERVENTIONS:
Drug: ramosetron 0.3 — The ramosetron 0.3 group receives ramosetron 0.3 mg at the end of surgery.
  Arms: ramosetron 0.3
Drug: ramosetron 0.45 — The ramosetron 0.45 group receives ramosetron 0.45 mg at the end of surgery.
  Arms: ramosetron 0.45
Drug: ramosetron 0.6 — The ramosetron 0.6 group receives ramosetron 0.6 mg at the end of surgery.
  Arms: ramosetron 0.6

SUMMARY:
Many patients receiving opioid based analgesia after gynecologic laparoscopic surgery experience postoperative nausea and vomiting (PONV) despite prophylaxis and treatment with HT3 receptor antagonists. Although a high dose of ramosetron can cause adverse effects such as headache or dizziness, the minimal effective dose of ramosetron in a high-risk patients is unknown. The aim of this study is to determine the effective dose of ramosetron for prophylaxis of PONV in a high-risk patients receiving intravenous opioid-based patient-controlled analgesia after gynecological laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* patient between 20 and 70 of age with ASA physical status Ⅰ-Ⅱ
* patient scheduled for elective gynecological laparoscopic surgery.

Exclusion Criteria:

* hepatorenal disease
* BMI > 35 kg/m2
* allergy to ramosetron
* gastrointestinal disease
* vomiting within 24h
* administration of antiemetics or opioids within 24h
* QT prolongation (QTc > 440ms)
* pregnant
* problem with communication

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2015-06-19 (Actual); Primary Completion 2016-02-06 (Actual); Study Completion 2016-02-06 (Actual)

PRIMARY OUTCOMES:
postoperative nausea and vomiting | within 48h after surgery
  incidence of nausea and vomiting during the first 48 h after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, 50 Yonsei-ro, Seodaemun-gu, Seoul, Seoul, South Korea